CLINICAL TRIAL: NCT03233750
Title: Preparing for High Acuity Events: Simulation-Based Stress Inoculation Training
Brief Title: Simulation-Based Stress Inoculation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170081-01H
Record Dates: First submitted 2017-07-13; First posted 2017-07-31 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Crew Resource Management, Healthcare

STUDY DESIGN:
Intervention Model Description: This is a cohort study, comparing two interventions aimed at decreasing stress responses during acute events, with a pre and a post intervention assessment.
Who Masked: Outcomes Assessor
Masking Description: Group assignment will be masked from the assessors of performance. Expert educators will score videotaped performances of the participants obtained pre and post intervention. Assessors will be blinded to group allocation as well as to whether the video they are scoring is of the pre or the post intervention scenario.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Inoculation Training (Experimental): Phase 1: Conceptualization / Educational Phase (60 minutes) Provision of preparatory information, to allow the participants to form accurate expectations regarding the stress environment and stress reactions.
  Phase 2: Skill Acquisition and Rehearsal (60 minutes) Development and practice of cognitive restructuring techniques and relaxing training to reduce anxiety and enhance the individual's capacity to respond effectively to stressful situations, in low stress conditions.
  Phase 3: Application of Coping Skills (180 minutes) Coping skills are applied in increasingly stressful conditions that approximate the real-world stressor environment.
  Interventions: Behavioral: Stress Inoculation Training
- Crisis Resource Management Training (Active Comparator): The CRM training targets the non-technical skills (e.g. behavioural and cognitive skills) required for effective teamwork during crisis situations. It focuses on communication, teamwork, situational awareness and leadership
  Interventions: Behavioral: Crisis Resource Management

INTERVENTIONS:
Behavioral: Stress Inoculation Training — see description in arm/group descriptions
  Arms: Stress Inoculation Training
Behavioral: Crisis Resource Management — During each scenario, facilitators identify performance gaps in either situation awareness, leadership, communication or resource allocations. During debriefing session, these are raised with the learner and their cognitive frames are identified and corrected as necessary.
  Arms: Crisis Resource Management Training

SUMMARY:
Previous research has shown that health professionals can experience stress responses during high acuity events such as trauma resuscitations. These stress responses can lead to impaired clinical performance. The goal of this proposed project is to adapt Stress Inoculation Training (SIT) to the healthcare setting. Stress Inoculation Training is a cognitive-behavioural approach to stress management that has proven effective in reducing stress and improving performance in domains outside of healthcare.

Thirty-two emergency medicine residents will be randomly divided into two groups. The SIT group will receive the simulation-based stress inoculation training. We will measure the effectiveness of the training by looking at reduction of stress levels and improvements in clinical performance in a pre-intervention and a post-intervention simulated trauma scenario. The control group will be exposed to the same simulation scenarios and pre/post intervention scenarios as the SIT group, but will not receive the stress inoculation training.

DETAILED DESCRIPTION:
Health care contains many stressors for health professionals, both chronic and acute. There is accumulating evidence that clinical performance can be significantly impaired by stress responses during acute events, both in the psychology and healthcare domains. Paramedics, medical residents and surgeons have all shown impaired performance when faced with high acuity situations that triggered subjective and physiological stress responses. Impairments have been observed in the ability to perform drug calculations, trauma and cardiac resuscitations, in technical skills, as well as on tasks that rely on memory recall. In some cases, the magnitude of the stress response has been associated with the degree of performance impairments. In many studies in which performance impairments have been observed, baseline levels of performance were acceptable, suggesting that these impairments are not due to a lack of relevant knowledge or skills required to provide patient care in these situations.

The findings of impaired performance with stress responses suggests that training for high acuity events needs to go beyond training that is oriented solely towards the acquisition of clinical skills and knowledge. Training needs to also include interventions aimed at developing the trainees' ability to cope with stressors and to minimize their personal stress responses. In the psychology, aviation and military domains, several approaches have been developed to optimize performance during stressful events. These can be categorized either as skills-based training (providing individuals or teams with the specific skills required during a crisis) or as stress management interventions (modifying the individual's appraisal of potentially stressful situations).

The implementation of skill based training, such as crisis resource management (CRM), has resulted in improved performance in team interactions. However, CRM-type of training requires that health professionals be able to remember those skills that were learned, yet memory recall is often impaired under stress. As for overlearning, it can lead to rigid approaches to problem solving, and is less likely to be efficient in dynamic situations that require flexibility in approaches and judgment. Therefore, educators also need to develop complementary approaches to train health professionals in recognizing stress responses and in managing and minimizing their emotional responses. Stress management approaches are focused on reducing the emotional and physiological response itself. The premise is that by reducing the stress response, the cognitive facilities (including recall of relevant knowledge and skills) required during a high acuity situation are more likely to remain intact.

Two important predictors of stress responses to high acuity events are individuals' coping styles and their cognitive appraisals of the situation. Task-oriented coping styles, as well as appraisals of perceived resources being equal to or above the perceived demands of a situation, are associated with lower stress responses in high acuity events. As such, stress management approaches focused on coping styles and cognitive structuring are likely to reduce the subjective and physiological stress responses of clinicians and trainees during high acuity events.

A promising method of reducing stress responses and performance impairments under acutely stressful conditions is stress inoculation training (SIT). This 3-phase cognitive-behavioural approach to stress management has proven effective in domains outside of healthcare. SIT has been found to be effective in reducing general state anxiety, performance anxiety (anxiety specific to the skills being addressed in the training), and in enhancing performance under stress. SIT appears to be effective when run with groups of 8-10 participants and it can be implemented successfully without an inordinate number of training sessions. Finally, the beneficial effects of the SIT can generalize to novel stress conditions and novel tasks, which is crucial for any applied area in which the conditions of real life environments are often dynamic, ambiguous and emergent.

The proposed study consists of the adaptation and evaluation of a simulation-based stress inoculation training (SIT) intervention for Emergency Medicine and Surgery residents during trauma rotations.

SPECIFIC AIMS AND HYPOTHESES The study hypothesis is that residents who have received the SIT intervention will have lower stress levels and higher performance levels during a post-intervention simulated trauma scenario than will residents in a control group.

SIGNIFICANCE During high acuity events, such as pre-hospital, trauma and cardiac resuscitations, patient care must be provided in conditions that can be noisy, chaotic, time pressured and with uncertainty. These conditions, and the urgent nature of the care required, are very unforgiving to gaps in recall, attention or decision-making. In these environments, research has shown that health professionals experience significant stress responses and that these stress responses can lead to impairments in memory, attention and clinical performance.

Adapting a proven stress training approach to healthcare has the possibility of significantly improving care to patients during high acuity events, both in terms of care during the high acuity component of care, as well as further along in the chain of care.

INNOVATION If, as predicted, the results of this study reveal that stress inoculation training is effective for preparing emergency medicine and surgery residents, in terms of reducing their stress levels and increasing their performance during simulated trauma resuscitation, this proposed study will be further developed for a multi-centre study with outcome measures of stress and performance during actual patient events.

In the development of the course content and scenarios for the SIT training in the context, a course manual will be produced. This manual will be shared with colleagues internationally, for the purposes of adapting and validating the course internationally and in a variety of clinical contexts.

APPROACH The proposed study of stress inoculation training (SIT) intervention will be for emergency medicine and surgery residents during trauma rotations. The adaptation of SIT to the trauma context will consist of a 3-phase training intervention, conducted over one 1/2 day session.

Phase 1: Conceptualization / Educational Phase (60 minutes) The goal of this phase is to help individuals gain a better understanding of the nature of stress and its effects. This phase will focus on the provision of preparatory information, to allow the participants to form accurate expectations regarding the stress environment and stress reaction that can occur during trauma cases. The goal is to provide the participants with a sense of predictability and control. This phase will consist of descriptions of the stressors encountered in the clinical setting, the provision of information about how these stressors might make the participants feel affect performance.

Phase 2: Skill Acquisition and Rehearsal (60 minutes) The objective of this phase is the development and practice of cognitive restructuring techniques and relaxing training to reduce anxiety and enhance the individual's capacity to respond effectively to stressful situations. The cognitive restructuring techniques will provide the participants with the skills to regulate negative emotions and distracting thoughts brought on by stressors. The relaxation training will provide the participants with the skills to enhance physiological control, such as awareness and control of muscle tension and breathing. The session will include mental imagery and visualization exercises to allow the participants to practice the skills in a low stress environment.

Phase 3: Application of Coping Skills (180 minutes) In this phase, the coping skills are applied in increasingly stressful conditions that approximate the real-world stressor environment. Participants will practice the cognitive restructuring and relaxation skills in a series of simulated trauma scenarios in which they will be exposed to increasing levels of stress in a gradual manner. All of the scenarios will be developed using a combination of computerized mannequin-based simulators and standardized patients (SP). The use of simulation modalities allows investigators to carefully manipulate the levels of stressors inherent in each scenario and to control for any extraneous factors beyond the intervention that could influence stress responses and performance.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine residents enrolled in post graduate training at the University of Toronto or the University of Ottawa

Exclusion Criteria:

* endocrine disease or medication that can affect cortisol levels or responses

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in scores on State-Trait Anxiety Inventory | prior to each scenairo as well as immediately at the end of each simulation scenario
  Subjective stress measure
Change in salivary cortisol levels | prior to each scenario, as well as 20 and 30 minutes after each scenario
  physiological indicator of stress

SECONDARY OUTCOMES:
Performance | Experts will review the videotapes of the scenarios within one month of data collection
  Expert scoring of clinical management of the scenario

CONTACTS AND LOCATIONS:
Overall Officials: Vicki LeBlanc, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
anonymized data shared on an individual basis